CLINICAL TRIAL: NCT05472402
Title: Feasibility and Acceptability of an Online Program to Promote Physical Activity Among Black Women
Acronym: LADIES Online
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gramercy Research Group (Other)
Responsible Party: Principal Investigator, Melicia Whitt-Glover, President & CEO, Gramercy Research Group
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: R21AG070657 (NIH)
Record Dates: First submitted 2022-07-18; First posted 2022-07-25 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Sedentary Behavior; Lack of Physical Activity; Physical Inactivity
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: The R21 phase will use 4 focus groups with 48 black women, and feedback from 12 expert advisors to modify content from our existing evidence-based PA curriculum for online implementation. - This phase has been completed.
  The R33 phase will use a randomized controlled trial design to implement a pilot study to evaluate the feasibility, acceptability, and impact on PA of the online PA curriculum.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LADIES online intervention (R33 phase) (Experimental): Participants will include 30 women who will be randomized to receive six (6) months of online group-based intervention sessions that teach participants how to increase physical activity levels.
  Interventions: Behavioral: LADIES online intervention (R33 phase)
- LADIES online control (R33 phase) (Placebo Comparator): Participants will include 30 women who will be randomized to receive self-guided materials that teach participants how to increase physical activity levels. Placebo comparator participants will receive their materials via the online platform.
  Interventions: Behavioral: LADIES online control (R33 phase)

INTERVENTIONS:
Behavioral: LADIES online intervention (R33 phase) — Participants will participate weekly online group sessions over 6 months. Participants will also receive access to written intervention materials, access to an online walking program, and access to weekly podcasts that are aligned with the intervention sessions and that support physical activity lessons with biblical scriptures.
  Other Names: LADIES online
  Arms: LADIES online intervention (R33 phase)
Behavioral: LADIES online control (R33 phase) — Participants will receive online access to a written self-guided curriculum that is self-paced and teaches participants how to increase physical activity. Participants will be encouraged to complete the self-guided curriculum within 6 months.
  Arms: LADIES online control (R33 phase)

SUMMARY:
This study will identify strategies for modifying a physical activity intervention, previously delivered in a face-to-face format, for online implementation.

DETAILED DESCRIPTION:
Research demonstrates the health-related benefits of participation in daily physical activity (PA), including prevention and treatment of chronic diseases. Despite this knowledge, the majority of US adults, particularly black women, do not achieve recommended levels of PA and, consequently, have higher rates of related chronic disease. An efficacy study led by the proposed Principal Investigator developed and tested an in person, 10-month group-based faith-integrated (FI) or secular (SEC) PA intervention, compared with a self-guided control (SG) for black women. Both FI and SEC were superior to SG for increasing daily steps after 10 months, and FI was superior to SG for increasing daily steps 12 months post intervention. Barriers to program participation noted by participants included childcare and work responsibilities and proximity to the group meeting location. The 2018 PA Guidelines Advisory Committee Scientific Report highlighted the need for effective strategies to promote PA, including internet-delivered interventions which have demonstrated strong evidence for effectiveness at increasing PA levels. Limited data exist regarding the efficacy of internet-delivered interventions in racial/ethnic minority groups. Online delivery of our evidence-based program may increase reach and address known barriers to PA program participation in black women. This project will explore strategies for adapting the program for web-based delivery of the existing curriculum. R21 phase aims are: Aim 1: Solicit input from individuals representative of the population of focus to inform the translation of the FI curriculum for online use; Aim 2: Use the knowledge gathered in Aim 1 to adapt existing FI and SG curricula for online use; Aim 3: Assess acceptability of the online curricula in an advisory group similar to the target population. Investigators will conduct focus groups with black women to understand factors that would influence online delivery of the curriculum. A 12-member advisory group will be convened to assist with developing materials/strategies to adapt the curriculum for online delivery. In an iterative approach where material is tested, refined, and retested until complete, investigators will engage the advisory group in feasibility testing of the online curriculum

ELIGIBILITY:
1. self-identified female
2. black/African American
3. > 18 years of age
4. self-reported low active (i.e., achieving < 150 minutes per week of moderate-to-vigorous physical activity)
5. no physical limitations or medical conditions that would be impacted by physical activity
6. own a smartphone or computer with reliable high speed internet access
7. able to speak and read English fluently; 8) potentially interested in participating in an online health intervention.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Self-reported female
Enrollment: 60 (Estimated)
Dates: Start 2022-05-22 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Daily step counts | Baseline and immediately post intervention
  Daily walking over 14 consecutive days
Bouts of moderate-to-vigorous physical activity | Baseline and immediately post intervention
  Daily bouts over 14 consecutive days using a wrist-worn accelerometer

SECONDARY OUTCOMES:
Sedentary behavior | Baseline and immediately post intervention
  Daily bouts over 14 consecutive days using a wrist-worn accelerometer
Self-reported physical activity | Baseline and immediately post intervention
  Participant reported using the 7-item self-administered modifided International Physical Activity Questionnaire
Clinical measures | Baseline and immediately post intervention
  Height, weight, seated blood pressure, waist circumference

CONTACTS AND LOCATIONS:
Overall Officials: Melicia Whitt-Glover, PhD, Principal Investigator — Gramercy Research Group; Robert Newton, PhD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Gramercy Research Group, Knightdale, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No